CLINICAL TRIAL: NCT03603795
Title: A Phase II Randomized Placebo-controlled Study to Assess the Impact on Outcome of Eltrombopag Administered to Elderly Patients with Acute Myeloid Leukemia Receiving Induction Chemotherapy
Brief Title: Study Impact on Outcome of Eltrombopag in Elderly Patients with Acute Myeloid Leukemia Receiving Induction Chemotherapy
Acronym: EPAG2015
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPAG 2015
Record Dates: First submitted 2018-04-20; First posted 2018-07-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — eltrombopag

STUDY DESIGN:
Intervention Model Description: Randomization between 2 arms
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Experimental): 55 patients will be randomized in the experimental arm A. If platelets counts < 100 x 10 Giga/L, patients will be treated with Eltrombopag 200 mg/day per os from day 11 of induction chemotherapy to platelets counts > 100 x 10 Giga/L or maximum to day 45. If platelets counts ≥ 100 x 10 Giga/L on day 11, the start of IP will be delayed until platelets < 100 x 10 Giga/L.
  Chemotherapy administration would be performed among standard practice:
  * Daunorubicin: 60 mg/m² D1 to D3
  * Cytarabine: 100 mg/m²/day, in a continuous 24h-IV infusion D1 to D7
  * Lomustine (CCNU): 200 mg/m² per os, at D1.
    200mg = 4 Tablets of 50 mg will be done more than 2 hours before Daunorubicin and cytarabine administrations, to avoid vomiting secondary to anthracycline administration.
  Investigational Product (IP) will be taken at the same time daily on an empty stomach 1 hour before or 2 hours after a meal or preferably no calcium or dairy products.
  Interventions: Drug: Eltrombopag
- B (Placebo Comparator): 55 patients will be randomized in the comparator arm B and will received: Placebo once daily from day 11 of induction chemotherapy to AML response evaluation or platelets count > 100 x 10 Giga/L (maximum day 45)
  Placebo 200mg = 4 Tablets of 50 mg will be done more than 2 hours before Daunorubicin and cytarabine administrations, to avoid vomiting secondary to anthracycline administration.
  Chemotherapy administration would be performed among standard practice:
  * Daunorubicin: 60 mg/m² D1 to D3
  * Cytarabine: 100 mg/m²/day, in a continuous 24h-IV infusion D1 to D7
  * Lomustine (CCNU): 200 mg/m² per os, at D1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag concomitant with induction chemotherapy in patient with AML
  Other Names: Arm Eltrombopag; Arm experimental A
  Arms: A
Drug: Placebo — Placebo concomitant with induction chemotherapy patients with AML
  Other Names: Arm placebo; Arm B
  Arms: B

SUMMARY:
Phase II randomized placebo-controlled study to assess the impact on outcome of Eltrombopag administered to elderly patients with Acute Myeloid Leukemia (AML) receiving induction chemotherapy. A phase II multicenter and randomized placebo-controlled study

DETAILED DESCRIPTION:
Subjects will be randomized 1:1 to receive Eltrombopag or matching placebo, in double blinded.

To compare overall survival rate at 12 months between the two arms, with or without 200 mg of Eltrombopag daily after induction chemotherapy

Arm A : Eltrombopag 200 mg (100 mg/day for east Asian heritage) once daily from day 11 of induction chemotherapy to AML response evaluation or platelets count > 100 x 10 Giga/L (maximum day 45)

Arm B : Placebo once daily from day 11 of induction chemotherapy to AML response evaluation or platelets count > 100 x 10 Giga/L. (maximum day 45)

ELIGIBILITY:
Inclusion Criteria

* 60 years of age.
* AML de novo, except AML 3 and AML 7.
* AML with no adverse cytogenetic according to Medical Research Council (MRC) 2010 classification.
* Subjects should be eligible for intensive chemotherapy by Daunorubicine, cytarabine, Lomustine.
* Eastern Cooperative Oncology Group (ECOG) < 3 (appendix 1).
* SORROR ≤ 3 (appendix 2).
* Adequate baseline organ function defined by the criteria below:

  * Total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) range except cases clearly not indicative of inadequate liver function
  * Alanine Aminotransferase (ALAT) and Aspartate Aminotransferase (ASAT) ≤ 3 x ULN
  * Creatinin ≤ 1.5 x ULN
* Adequate cardiac function with Left Ventricular Ejection fraction (LVEF) ≥50%
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Women will be menopausal to be enrolled
* The patient must give written (personally signed and dated) informed consent before completing any study-related procedure which means assessment or evaluation that would not form part of the normal medical care of the patient and before the start of induction chemotherapy.
* Affiliated to the French Social Security (Health Insurance).

Exclusion criteria

* Subjects with a diagnosis of acute promyelocytic (M3) or megakaryocytic leukemia (M7).
* AML with adverse cytogenetic according to the MRC 2010 classification.
* AML secondary to Myelodysplastic syndrome (MDS), Myeloproliferative neoplasm (MPN)
* Clinical symptoms suggesting active central nervous system leukemia, or presence of extramedullary AML.
* Previous exposure to anthracycline.
* Previous AML treatment other than hydroxyurea.
* Treatment with an investigational drug within 30 days or 5 half-life whichever is longer, preceding the first dose of study medication.
* History of thromboembolic event or other condition requiring ongoing use of anticoagulation either with warfarin or low molecular-weight heparin.
* History of another malignancy within the past three years except basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Pre-existing cardiovascular disease (including congestive heart failure, New York Heart Association (NYHA) Grade III/IV), or arrhythmia known to increase the risk of thromboembolic events (e.g. atrial fibrillation), or subjects with a QTc >450 msec (QTc >480 msec for subjects with Bundle Branch Block).
* Patient requiring platelets transfusion with platelets > 10 x 10 Giga/L, for whatever reason.
* History of treatment with romiplostim or other Thrombopoietin receptor (TPO-R) agonists.
* Uncontrolled active infection.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would place the participant at an unacceptable risk or prevent them from giving informed consent.
* Known active HIV, Hepatitis B or C infection.
* Pregnancy or breastfeeding.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-10-11 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Overal survival rate | 12 months after beginning treatment
  overall survival rate at month 12 (year 1) between the two arms, with or without 200 mg of Eltrombopag daily after induction chemotherapy.

SECONDARY OUTCOMES:
Response rate (CR and CRi) at day 45 | At day 45
Leukemia Free Survival at month 12 (one year) | 12 months after beginning treatment
  relapse measurement before month 12
Long-term survival | 2, 3 and 5 years after first treatment administration
  Overall survival at 2, 3 and 5 years
Percentage of patients with platelets count > 100 Giga/L at day 45 | At day 45
  platelets count >100 Giga/L
Time to platelet transfusion independence | platelets count daily from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  More than 3 days with platelets count ≥ 10 Giga/L

OTHER OUTCOMES:
Number of accident haemorrhage events ≥ grade 3 | Until day 45
  All accident haemorrhage event ≥ grade 3
Number of days with platelets count <10 Giga/L | from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  Daily measurement of platelets count
Number of platelets transfusion | from baseline to the end of induction (day 45)
Time to platelets count > 100 Giga/L | from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  Daily measurement of platelets count
Time to peripheral blood polymorphonuclear neutrophils (PMN) counts > 0.5 G/L | from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  Daily measurement of peripheral blood PMN count
Time to haemoglobin counts > 8 g/dl | from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  Daily measurement of haemoglobin count
Time to red blood cells transfusion independence | from baseline to the end of induction (day 45) and then at day 60, day 90, monthly until year 1 and finally at year 2, year 3 and year 5
  Daily measurement of Red blood cells count and transfusion monitoring
Eltrombopag-Emergent Adverse Events | Until day 90
  Incidence and severity of Eltrombopag-Emergent Adverse Events utilizing National Cancer Institute - Common Terminology Criteria (NCI-CTC) criteria v4.03
Evaluation of quality of life | At baseline and at the end of induction (maximum up to day 45)
  EORTC Quality of Life Questionnaire - Core Questionnaire (QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud PIGNEUX, MD PD, Principal Investigator — French Innovative Leukemia Organization (FILO)
Locations (15):
- France (15):
  - CHU ANGERS - Maladies du sang, Angers
  - CH de la Côte Basque - Hématologie, Bayonne
  - CHU Estaing, Clermont-Ferrand
  - CHU Grenoble - Hématologie Clinique, Grenoble
  - Institut Paoli-Calmettes - Hématologie 2, Marseille
  - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - HOPITAL E. MULLER - Hématologie, Mulhouse
  - CHU HOTEL DIEU - Hématologie Clinique, Nantes
  - CHU Caremeau, Nîmes
  - CHU La Milétrie - Hématologie Clinique, Poitiers
  - CHU Pontchaillou, Rennes
  - CHU Hautepierre - Hématologie, Strasbourg
  - Institut Universitaire du Cancer de Toulouse Oncopole - Service d'Hématologie, Toulouse
  - Sponsor FILO, Tours
  - CHU de Brabois, Vandœuvre-lès-Nancy

REFERENCES:
- See also: FILO internet site — http://www.filo-leucemie.org